CLINICAL TRIAL: NCT05512715
Title: A Randomized Controlled Clinical Trial on the Effectiveness of Lithium in Comparison to Carbimazole as a Bridging Therapy Prior to Radioactive Iodine for Hyperthyroidism
Brief Title: LIthium as Bridging thErapy Prior to Radioactiveiodine in hyperThYroidism
Acronym: LIBERTY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JEP-2020-763
Record Dates: First submitted 2022-08-20; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-07

CONDITIONS: Hyperthyroidism/Thyrotoxicosis
MeSH Terms: conditions — Hyperthyroidism; Thyrotoxicosis

STUDY DESIGN:
Intervention Model Description: randomised into lithium or carbimazole arms in a 1:1 ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lithium (Active Comparator): Tablet Lithium Carbonate 300mg daily for 2 months
  Interventions: Procedure: radioactive iodine
- Carbimazole (Active Comparator): Tablet Carbimazole 10mg daily for 2 months
  Interventions: Procedure: radioactive iodine

INTERVENTIONS:
Procedure: radioactive iodine — radioactive iodine 15mci

SUMMARY:
A prospective randomised controlled open label, single centre study. subjects will be randomised into lithium or carbimazole arms in a 1:1 ratio. Lithium arm will receive tab Lithium Carbonate 300mg daily while Carbimazole arm will receive tab Carbimazole 10mg daily for a duration of two months prior to radioactive iodine treatment. Changes in the thyroid hormone levels at 2 months of treatment and at months 1,3 and 6 following radioactive iodine will be evaluated.

DETAILED DESCRIPTION:
This is a prospective randomized, open label, single center interventional study comparing the effectiveness of lithium versus carbimazole in lowering the thyroid hormone levels in patients undergoing radioactive iodine. Patients will be randomized into lithium or carbimazole arms in a 1:1 ratio. Patients will receive either lithium carbonate 300mg once daily or carbimazole 10mg once daily, which is the current standard therapy. The necessary precautions will be given with regards to the study drugs. Patients will be on the above treatment for a duration of 2 months and carbimazole will be stopped 3 days prior to radioactive iodine treatment whereas lithium will be discontinued on day 3 post RAI as per usual practice. RAI will be administered at a fixed dose of 15mCi in both groups.

Antithyroid drug (ie. Methimazole or carbimazole) is restarted if needed (in symptomatic patients with FT4 of more than 40 pmol/L) at least a week after radioactive iodine and titrated as per standard treatment protocol. Patients are declared to be cured at the end of 6 months based on thyroid function test and requirement of treatment either with thyroxine or antithyroid drug.

Block randomization method will be utilised to randomize subjects into the two groups by selecting treatment arm from a box consisting of 8 options (4 lithium and 4 carbimazole). Once the box is empty, it will replenished by the same 8 options.

Patients who are able to comply with the requirement of radioiodine therapy and consented to participate in this trial will be given appropriate counselling. These patients will be screened for inclusion and exclusion criteria. A written informed consent will be obtained and patients will then be recruited into this study.

Once recruited, history, physical examination including baseline eye examination for possible Thyroid Eye Disease (TED) will be carried out. TED as defined according to the presence of eye signs in categories 2-6 of the NOSPECS classification and determined clinical activity score of thyroid eye disease according to EUGOGO criteria. Patients will be then assessed for baseline thyroid function test (TFT), renal profile (RP) and liver function test (LFT) during screening. Patients will receive either lithium carbonate 300mg once daily or carbimazole 10mg once daily, which is the current standard therapy. The necessary precautions will be given with regards to the study drugs. Patients will be enquired of any possible side effects during the clinic visits. Lithium levels will be checked at week 1 and at the end of 2 months of initiation (refer study flow chart). If patient develops intolerable side effects or the lithium level exceeded therapeutic range, the confounding drug will be stopped and patient will be managed accordingly. The patient will subsequently be withdrawn from the study. It is important to note that the lithium dose used in this study is of low dose, hence the side effects risks anticipated would be low. Current waiting period in PPUKM is about 2months. Patients will be on the above treatment for a duration of 2 months and carbimazole will be stopped 3 days prior to radioactive iodine treatment. RAI will be administered at a fixed dose of 15mCi in both groups. Bloods will be drawn for TFT, RP, LFT and lithium level on the RAI day. Lithium will be discontinued on day 3 post RAI. The timeline for stopping both the carbimazole and lithium are as per clinical practice guidelines. Patients will be followed up at months 1, 3 and 6 post RAI with TFT during each visit.

All adult patients who are 18 years and above with hyperthyroidism either newly diagnosed or relapse disease secondary to Graves' Disease, toxic multinodular goitre and toxic adenoma who are planned for radioactive iodine therapy as a definitive treatment will be included in this study. The study period is from 10/1/2021 till 31/5/2022 at Pusat Perubatan Universiti Kebangsaan Malaysia.

ELIGIBILITY:
Inclusion Criteria:

Adult patients aged 18 years old and above with thyrotoxicosis who have been planned for definitive radioactive iodine:

* consented for radioactive iodine as a definitive treatment
* able to comply with requirement of radioactive iodine treatment
* FT4 level below 40pmol/L

Exclusion Criteria:

* pregnancy or lactating mother
* moderate to severe and active thyroid eye disease based on EUGOGO criteria, requires steroid cover
* renal impairment, egfr <45mls/min (stage 3b)
* underlying activity malignancy
* underlying active schizophrenia or bipolar disorder
* patients on medication that may interact with lithium (refer appendix)
* patients on medications that may interfere with radioactive iodine effectiveness such as amiodarone and less than a month of intravenous contrast medium
* previous radioactive iodine less than 6 months
* previous history of adverse effect following exposure to lithium or carbimazole
* thyroid carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
proportion of cure at 6months | 6 months
  to assess the proportion of cure at 6 months of radioactive iodine between those who were pre-treated with lithium vs carbimazole

SECONDARY OUTCOMES:
change in serum thyroid hormone | 2 months
  to assess the change in serum thyroid hormone levels following two months of lithium versus carbimazole therapy prior to the administration of radioactive iodine

CONTACTS AND LOCATIONS:
Overall Officials: Norlela Sukor, Principal Investigator — Hospital Canselor Tuanku Muhriz
Locations (1):
- Hospital Canselor Tuanku Muhriz, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT05512715/Prot_000.pdf